CLINICAL TRIAL: NCT01514630
Title: Creatine as a Treatment Option for Depression in Methamphetamine Using Females
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Perry Renshaw (Other)
Responsible Party: Sponsor-Investigator, Perry Renshaw, Professor of Psychiatry, University of Utah
Organization: University of Utah (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 60398
Record Dates: First submitted 2012-01-12; First posted 2012-01-23 (Estimated); Results first posted 2015-06-29 (Estimated); Last update posted 2015-06-29 (Estimated); Status verified 2015-06

CONDITIONS: Depression; Substance Abuse; Substance Use; Neuroimaging; Dual Diagnosis
MeSH Terms: conditions — Depression; Substance-Related Disorders | interventions — Creatine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Creatine monohydrate (Experimental): 14 female depressed methamphetamine users received 5 grams of creatine monohydrate daily for eight weeks.
  Interventions: Drug: Creatine monohydrate

INTERVENTIONS:
Drug: Creatine monohydrate — Five grams of creatine monohydrate will be administered for eight weeks.

SUMMARY:
Methamphetamine (MA) is a psychostimulant drug with high abuse potential. MA can be smoked, snorted, injected or ingested orally to produce a release of high levels of dopamine into the brain and reduction of dopamine uptake. Its use results in feelings of pleasure, increased energy, and greater alertness lasting up to 12 hours. In 2010, the National Survey on Drug Use and Health reported that 353,000 Americans aged 12 or older reported being current MA users. Over the past decade MA use rates have fluctuated with current use rates on the decline; however, importantly, even though overall use rates are declining, use rates among males and females are approaching equal proportions. This use rate pattern is unlike other drugs of abuse, which typically demonstrate males using more than females. In some states, more females than males consider MA as their drug of choice. Namely, in a 2010 report in the state of Utah, more females were diagnosed with MA as a primary substance of abuse than males upon admission to treatment.

Depression and MA use are highly comorbid. The relationship between MA use and depression is likely bidirectional, with MA use causing changes in mood and being used as a self-medicating behavior to reduce symptoms of depression. Several studies have shown that depression rates are higher in MA-using females compared to their male counterparts. It is likely that neurobiological and psychosocial mechanisms contribute to increased incidence of depressive symptoms in females.

No clear treatment model exists to suggest how the comorbidity of depression and MA use is best managed. In studies of antidepressants for treatment of MA withdrawal and dependence, findings have suggested that antidepressants are ineffective for treating depressive symptoms.

Creatine is an organic acid occurring naturally in vertebrates, where it takes part in energy homeostasis in tissues with fluctuating energy demands. Exogenous creatine has been shown to increase brain concentrations of PCr. Neuroimaging studies of creatine have shown increased brain phosphocreatine (PCr) content with creatine administration. Therefore, we hypothesize that oral creatine administration will increase PCr levels and reduce depressive symptoms in a sample of depressed female MA users. This hypothesis will be tested by a within subjects design by giving depressed MA using females oral creatine for eight weeks and measuring PCr pre- and post-treatment with magnetic resonance spectroscopy. Moreover, depressive symptoms will be measured by administration of the Hamilton Depression Rating Scale twice weekly during the course of creatine treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Female gender, ages 18-64 years inclusive
2. Diagnosis of MA dependence or abuse within the past 12 months, with MA preferred drug of abuse, identified by the SCID-I-RV
3. Current diagnosis of Major Depressive Disorder identified by the SCID-I-RV
4. Current HAM-D17 score of > 15

Exclusion Criteria:

1. Diagnosis of bipolar disorder, schizophrenia, or schizoaffective disorder, identified by the SCID-I-RV
2. History of or current diagnosis of renal disease, such as chronic renal failure, acute renal failure or end stage renal disease
3. Diabetes type I or II
4. Colitis or diverticulitis
5. Seizure disorder
6. Current serious suicide risk identified by the Columbia Severity Suicide Rating Severity
7. Current treatment with an antipsychotic, mood stabilizer, or antidepressant
8. Positive HIV test
9. Active Hepatitis C
10. Contraindication to magnetic resonance scan

Ages: 13 Years to 64 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 14 (Actual)
Dates: Start 2013-01; Primary Completion 2014-12 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tracy Hellem, RN, Principal Investigator — The College of Nursing & Brain Institute, University of Utah; Perry Renshaw, MD, PhD, MBA, Study Director — Department of Psychiatry, University of Utah
Locations (1):
- The Brain Institute of the University of Utah, Salt Lake City, Utah, United States

REFERENCES:
- [Derived] Hellem TL, Sung YH, Shi XF, Pett MA, Latendresse G, Morgan J, Huber RS, Kuykendall D, Lundberg KJ, Renshaw PF. Creatine as a Novel Treatment for Depression in Females Using Methamphetamine: A Pilot Study. J Dual Diagn. 2015;11(3-4):189-202. doi: 10.1080/15504263.2015.1100471. PMID 26457568

RESULTS

PARTICIPANT FLOW:
Groups:
- Creatine Monohydrate: 14 female depressed methamphetamine users received 5 grams of creatine monohydrate daily for eight weeks. Participants were seen twice weekly after creatine was initiated. All participants met SCID-I/P criteria for lifetime methamphetamine dependence or for current methamphetamine dependence. After consent was obtained, the principal investigator administered the SCID-I/P and HAMD, and if a female met SCID-I/P criteria and scored > 15 on the HAMD, the following additional screening data were collected: Beck Anxiety Inventory, C-SSRS , vital signs, concomitant medications, self-report drug use over the past 48 hours for cigarettes, alcohol, cocaine, methamphetamine, marijuana, heroin and prescription controlled substances, urine drug screen for methamphetamine, opiates, benzodiazepines, marijuana and cocaine, pregnancy testing and attendance in outpatient treatment and/or 12 step programs.
Period: Overall Study
Arm/Group | Creatine Monohydrate
Started | 14
Completed | 11
Not Completed | 3

BASELINE CHARACTERISTICS:
Groups:
- Creatine Monohydrate: 14 female depressed methamphetamine users will receive 5 grams of creatine monohydrate daily for eight weeks.
  Creatine monohydrate: Five grams of creatine monohydrate will be administered for eight weeks.
Arm/Group | Creatine Monohydrate
Number analyzed (Participants) | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 14
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.4 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 14

OUTCOME MEASURES:

1. Primary Outcome: HAMD Rating Scores
Description: Eight weeks of oral creatine supplementation will result in improvements in Hamilton Depression Rating Scale (HAMD) in female methamphetamine users. HAMD scoring is based on 17 items. Minimum score is 0 and maximum 52. A score of 0-7 is considered to be normal. Scores of 20 or higher indicate moderate or severe depression.
  0-7 = Normal 8-13 = Mild Depression 14-18 = Moderate Depression 19-22 = Severe Depression
  ≥ 23 = Very Severe Depression
Time Frame: Over the course of eight weeks. Depression rating scores will be measured weekly for eight weeks for each subject enrolled.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Creatine Monohydrate
Number analyzed (Participants) | 11
Units on a scale
  Baseline | 16.86 (3.40)
  week 2 | 10.71 (4.75)
  week 3 | 9.81 (4.45)
  week 4 | 7.33 (2.74)
  week 5 | 8.35 (4.12)
  week 6 | 7.73 (3.88)
  week 7 | 6.28 (5.07)
  week 8 | 7.36 (4.59)

ADVERSE EVENTS:
Arm/Group | Creatine Monohydrate
Serious Adverse Events (participants affected / at risk) | 0/14
Other Adverse Events (participants affected / at risk) | 14/14
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Creatine Monohydrate (N=14)
Cold and flu symptoms (General disorders) | 10
Indigestion (Gastrointestinal disorders) | 1
Polydipsia (General disorders) | 1
Headache (General disorders) | 1
Swelling in Hands (General disorders) | 1
Diarrhea (Gastrointestinal disorders) | 4
Stomach Discomfort (Gastrointestinal disorders) | 3
Numbness and Tingling in hands (General disorders) | 1
Muscle Cramps (General disorders) | 2
Lightheaded (General disorders) | 1
Nausea (General disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No